CLINICAL TRIAL: NCT06752148
Title: Quantitative Measurement of Brain State and Neurofeedback Intervention Techniques for the Treatment of Perioperative Neurocognitive Disorders in Elderly Patients
Brief Title: Quantitative Neurofeedback Techniques for Treating Perioperative Cognitive Disorders in Elderly Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2022-JKCS-20
Record Dates: First submitted 2024-08-03; First posted 2024-12-30 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Emergence Delirium; Perioperative Neurocognitive Disorder
Keywords: perioperative neurocognitive disorder; neurofeedback intervention training; elderly patients; quantitative measurement of brain
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Subjects should undergo at least 2 consecutive weeks of uninterrupted closed-loop neurofeedback training prior to surgery. During the training cycle, subjects can train "Digital Meditation" (15-20 minutes) + "Idea Magic Ball" game (5-15 minutes) at least once a day in the morning and once in the afternoon, and then choose whether or not to play the "Chase Training" and "Concentration Training" games. The "Chase Training" and "Concentration Training" games should be played at your own choice. During the cycle, you need to perform "sleep induction" training once a night before going to bed (20-40 minutes), and complete the cumulative ≥14 hours of training (the length of time recorded by the APP) before the surgery. The total number of hours of training should be ≥14 before the surgery (APP records the number of hours of training).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Medical staff and outcome assessors were blinded to the fact that volunteers were responsible for obtaining the randomisation number, preparing the intervention equipment, and training in its use, and that patient follow-up, and assessment of relevant outcomes, were carried out by a trained investigator (anaesthetist), who was not involved in anaesthesia or perioperative management; medical staff and other investigators, except volunteers, were not aware of the subgroups; and the study was not blinded to the subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects should undergo at least 2 consecutive weeks of uninterrupted closed-loop neurofeedback training prior to surgery. During the training cycle, subjects can train "Digital Meditation" (15-20 minutes) + "Idea Magic Ball" game (5-15 minutes) at least once a day in the morning and once in the afternoon, and then choose whether or not to play the "Chase Training" and "Concentration Training" games. The "Chase Training" and "Concentration Training" games should be played at your own choice. During the cycle, you need to perform "sleep induction" training once a night before going to bed (20-40 minutes), and complete the cumulative ≥14 hours of training (the length of time recorded by the APP) before the surgery. The total number of hours of training should be ≥14 before the surgery (APP records the number of hours of training).
  Interventions: Combination Product: neurofeedback intervention training game
- Control Group (No Intervention): Control subjects lived a normal life before the operation.

INTERVENTIONS:
Combination Product: neurofeedback intervention training game — 1. Issuance of training equipment and training in its use: For subjects randomly assigned to the intervention group, a volunteer who has received adequate training in the use of the equipment will issue the EEG monitoring electrodes (model: HXD-1) and paired PADs, and will provide an activated account for the use of the subject only and training in its use. Subjects will be provided with a short tutorial on how to use the APP, which is very user-friendly and suitable for elderly novices. An initial training session will consist of 3 training components and will be completed with a volunteer.
  2. Training programme and supervision: The closed-loop neurofeedback training will consist of 3 parts, namely "Digital Meditation", "Brain Training" and "Sleep Induction". The "brain training" will consist of three games: "Idea Chase", "Idea Magic Ball" and "Focused Archery". The control subjects lived a normal life before the surgery, and all subjects underwent the surgery as planned.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if quantitative measurement of brain and neurofeedback intervention techniques works to prevent perioperative neurocognitive deficits in elderly oncology patients who are to undergo elective major surgery. The main questions it aims to answer are:

* Can neurofeedback intervention training reduce the incidence of postoperative delirium in elderly oncology patients? Researchers will compare the incidence of postoperative delirium in elderly oncology patients after training in neurofeedback intervention with those after living a normal life, to see if training in neurofeedback intervention before surgery is effective in preventing the development of postoperative delirium.

Participants will:

* Take neurocognitive feedback intervention training for 14 days prior to surgery (recommended to be used for at least 1 hour per day for a cumulative preoperative use of 14 hours).

  * Received preoperative and postoperative assessments of cognitive function by a third-party researcher, as well as daily delirium assessments for 7 days postoperatively.

    * The subjects in the control group lived a normal life every day before the operation, and the rest of the measures were the same as those in the intervention group.

DETAILED DESCRIPTION:
* Study design: The present study is a randomized controlled clinical trial in which subjects were screened on the basis of inclusion and exclusion criteria and were randomised into the following control group (n=195) and intervention group (n=195) in a ratio of 1:1.

  ②Participants: A total of 390 patients will be enrolled in this study, all of whom will be elderly patients undergoing elective surgery at the Cancer Hospital of the Chinese Academy of Medical Sciences (CAMS)/Beijing Chaoyang Hospital (BCH)/Xuanwu Hospital (Xuanwu Hospital). The main inclusion and exclusion criteria are listed below: Inclusion criteria：
  1. Patients undergoing elective major surgery (colorectal, pancreatic-gastric, hepatobiliary, thoracic, gynaecological and urological) under general anaesthesia;
  2. Expected duration of surgery >2 hours;
  3. Age ≥65 years; Exclusion criteria：

  <!-- -->

  1. refused to participate in this study;
  2. preoperative MMSE score <26 or if the patient's educational level was lower than high school, MMSE <24 and active depressive state (GDS-15 score >9);
  3. underwent neurosurgery or the surgery itself interfered with the patient's postoperative communicative communication (e.g., tracheotomy);
  4. severe organ dysfunction;
  5. underwent cardiac surgery, (e) Undergoing cardiac surgery, neurosurgery, or neurosurgery; (f) ASA classification IV or higher.

     ③Sample size，Randomisation and blinding： Referring to the results of the previous study, assuming that the incidence of POD in patients in the intervention group was 8% and the incidence of POD in patients in the control group was 18%, according to the statistical efficacy of 80%, the test level of unilateral 0.025, and the test of superiority using the PASS 15 software Tests for Two Proportions, the calculation of the intervention group: the control group = 1:1, each of the two groups needed 177 cases. A total of 354 cases. Considering the dropout rate of about 10% during the clinical trial, the minimum number of cases in the intervention group and the control group was 195 cases, and it was estimated that a total of 390 cases were needed.

     Recruitment and informed consent：Patients will be screened by dedicated investigators at designated surgical clinics and anaesthesia clinics, as illustrated in the screening process. Surgeons and anaesthesiologists will conduct prospective screening based on the inclusion/exclusion criteria specified in the protocol, and the investigator will be required to keep a screening log, and patients who meet the inclusion criteria will need to be recorded in the screening log, which will be filled in by the investigator, and a written informed consent will be signed by the investigator with the patient's consent. If the inclusion criteria are met but patients are not recruited, the reasons for not enrolling in the trial need to be recorded in the screening log.

     Randomisation and blinding: The study was grouped using stratified block randomisation with known risk factors for POD: age ≥80 years, dementia and poor physical condition, stratified by sex, age 65-79 years, 80 years and over and ASA grade 1/2/3, and then block randomised by generating random numbers in a 1:1 ratio through a 24-hour online central randomisation system.

     Medical staff and outcome assessors were blinded to the fact that volunteers were responsible for obtaining the randomisation number, preparing the intervention equipment, and training in its use, and that patient follow-up, and assessment of relevant outcomes, were carried out by a trained investigator (anaesthetist), who was not involved in anaesthesia or perioperative management; medical staff and other investigators, except volunteers, were not aware of the subgroups; and the study was not blinded to the subjects.
     * Withdrawal or termination of research: The investigator should facilitate the completion of the entire study for each subject whenever possible. Subjects may withdraw from this study for any reason.

       1. Serious adverse events: e.g., the patient has difficulty tolerating the neurofeedback intervention training and has adverse reactions such as nausea, dizziness, headache, etc.; the patient is allergic to the electrodes and related materials, and has difficulty tolerating the brain state testing and neurofeedback intervention training;
       2. Subjects request to withdraw from the study;
       3. The investigator decides whether the subject withdraws from the study on a case-by-case basis; Once a subject withdraws from the study, the study should notify the Team Leader as soon as possible and make best efforts to complete the pre-withdrawal assessment. All subjects who withdraw from the study due to an adverse event should be followed up until the adverse event has completely resolved, after the investigator has judged that the adverse event is in a stable phase or lost to follow-up, and for all subjects who withdraw from the study, the date of withdrawal and the reason for withdrawal, etc., should be recorded in detail on the CRF form.

     Subjects could terminate participation in the study at any time and would not be biased in subsequent treatment. If a subject terminates the study, the reason is documented with the CRF form. If the subject terminates the intervention training early and asks to withdraw, the investigator is required to make every effort to complete the remaining study visits, as shown in the study flow chart, including visits 1 day preoperatively, within 7 days postoperatively, and 30 days postoperatively.

     If the subject asks to withdraw and refuses the functional brain status test and questionnaire assessment, the investigator should explain the importance of remaining in the study for the trial follow-up, and if the patient still refuses, allow routine follow-up data such as the occurrence of postoperative POD, postoperative complications, postoperative hospital stay, and total hospitalisation costs to be used for the trial purposes, as well as allow the use of existing collected data.

     If subjects have less than the recommended length of training, less than 2 hours of surgery, or less than 7 days of postoperative hospitalisation after enrolment resulting in partial loss of study data, the investigator must still make every effort to complete the remainder of the study visit, at which point the patient is still within the trial and data collection and analysis can still be performed.
     * data management （a）The investigator enters the data into the EDC system in a timely, complete and correct manner based on the subject's original observations; （b）Supervisors monitor that tests are conducted in accordance with the test programme and that data are entered in a timely manner; （c）The EDC system completes data entry and verification as required, and then files and maintains it as required.

       * statistical analysis （a）Descriptive analysis of demographic and clinical characteristics: Measurements were expressed as mean and standard deviation (X±SD) if they obeyed normal distribution, or median (M) and interquartile spacing if they were skewed. For comparison between the two groups, Student-t test was used if the variables obeyed normal distribution, and Mann-Whitney U test was used if they obeyed skewed distribution. Count data were expressed as frequencies and percentages, and comparisons between groups were made using the χ2 test or Fisher's exact probability method.

         （b）Efficacy analysis: POD will be identified by CAM on postoperative days 0-7, and POD-positive patients will be followed until the patient recovers from delirium. The incidence of POD in the intervention and control groups will be compared using the χ2 test of superiority, and differences in STAI, PSQI and MMSE between groups will be compared using the Student-t test or the χ2 test.
         * Quality Control and Quality Assurance

           1. Training of researchers and medical personnel: the research programme should be explained in detail to the researchers and medical personnel before the commencement of the study, and the research programme must be strictly observed during the study period, and the researchers must first receive the training of subjects before they can take part in the study; the researchers should carry out the test in strict accordance with the research programme, and fill in the case report form completely, in detail and accurately, and all the observed results and abnormal findings in the clinical trial should be carefully verified and recorded in time to ensure the reliability of the data; all the instruments and equipment used in the test should be of strict quality standards and ensure normal operation; when summarizing and analyzing the results of the clinical trial, standardized standards should be adopted to ensure that the data is reliable. All the observed results and abnormal findings in the clinical trial should be verified and recorded in a timely and serious manner to ensure the reliability of the data; all the instruments and equipments used for the various checking items in the trial should be of strict quality standards and ensure normal operation; when summarising and analysing the results of the clinical trial, standardised methods of statistical analysis must be adopted and personnel familiar with biostatistics should be invited to take part in the trial; All kinds of conclusions of clinical trials must be derived from original data.
           2. Supervision during the study: The designated project supervisor will carry out project supervision of the study, the purpose of which is to ensure that the implementation of the study, data recording and analysis are carried out in accordance with the study protocol and relevant regulations. The supervisor will carry out supervision of the study in accordance with the Supervision Plan, which includes on-site supervision visits and remote supervision.

              * ethical requirements： （a）Clinical trials are conducted in accordance with the Declaration of Helsinki and relevant Chinese clinical trial management norms. Prior to the commencement of the trial, the trial protocol was approved by the Clinical Research Ethics Committee before the clinical trial could be implemented; （b）Before each patient is enrolled in this study, it is the responsibility of the investigating physician to provide a complete and comprehensive description of the purpose, procedures, and possible risks of this study in written text. Patients will be made aware of their right to withdraw from the study at any time. Each patient must be given a copy of the informed consent form prior to enrolment and it is the responsibility of the research physician to obtain informed consent before each patient enters the study.The informed consent form is retained as clinical trial documentation for review. For the purposes of this trial, the patient and his/her authorised representative under anaesthesia should be informed of the above and sign the informed consent and power of attorney prior to the procedure. (The power of attorney is in our standardised version).

                （c）The results of the study will be published in the form of a paper, but all personal information of the participants should be kept confidential.

                ⑨Termination of the study: In the event of a trial-related death during the study, the study will be terminated early and reported promptly to the Ethics Committee. Restarting the study will require ethics committee approval; After completing patient enrolment and data collection under normal circumstances, the study of a clinical trial may be closed with the consent of the principal investigator.
                * Custody of documents EDC data is kept for at least 5 years as required by GCP.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective major surgery (colorectal, pancreatic-gastric, hepatobiliary, thoracic, gynaecological and urological) under general anaesthesia;
* Expected duration of surgery >2 hours;
* Age ≥65 years;

Exclusion Criteria:

* refused to participate in this study;
* preoperative MMSE score <26 or if the patient's educational level was lower than high school, MMSE <24 and active depressive state (GDS-15 score >9);
* underwent neurosurgery or the surgery itself interfered with the patient's postoperative communicative communication (e.g., tracheotomy);
* severe organ dysfunction;
* underwent cardiac surgery, (e) Undergoing cardiac surgery, neurosurgery, or neurosurgery;
* ASA classification IV or higher.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 7 days after surgery
  On postoperative days 1-7, the investigator assessed subjects for CAM daily from 8:00 am-12:00 pm and 14:00 pm-18:00 pm.

SECONDARY OUTCOMES:
Number of occurrences of delirium | 7 days after surgery
  Researchers recorded the number of times subjects experienced delirium in the 7 days following surgery.
Severity of POD | 7 days after surgery
  For subjects diagnosed with postoperative delirium within 7 days of surgery, the severity of delirium was assessed using Confusion Assessment Method-Severity Short Form. This scale includes a total of 4 items, with a scoring range of 0-7 points, where 0 points indicate no delirium, 1 point indicates mild delirium, 2 points indicate moderate delirium, and 3-7 points indicate severe delirium.
Type of POD | 7 days after surgery
  For subjects diagnosed with postoperative delirium within 7 days after surgery, the type of delirium is determined based on their presentation. Hyperactive delirium is characterized by alertness, agitation, and increased psychomotor activity; hypoactive delirium is characterized by apathy, drowsiness, and reduced psychomotor activity; mixed delirium is characterized by alternating features of hyperactivity and hypoactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zheng, MD, Principal Investigator — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT06752148/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT06752148/ICF_001.pdf